CLINICAL TRIAL: NCT06562569
Title: Stimulating the Vagus Nerve to Improve Gait in Veterans With Parkinson's Disease
Brief Title: Non-invasive VNS for PD Gait
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E5133-P
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
Keywords: vagal nerve stimulation; gait; neuromodulation; Freezing of gait; Veteran
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Veterans will be randomized to one of two groups that will receive vagal nerve stimulation
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Vagal nerve stimulation at an intensity under 10 units. Participants will self-administered at this intensity for 2 minutes each day over 4 weeks.
  Interventions: Device: non-invasive cervical vagal nerve stimulation ncVNS
- Group 2 (Experimental): Vagal nerve stimulation at the highest intensity tolerated by the participant. Participants will self-administered at this intensity for 12 minutes each day over 4 weeks.
  Interventions: Device: non-invasive cervical vagal nerve stimulation ncVNS
- Group 3 (No Intervention): This group will not receive any stimulation. Participants will receive their treatment as usual.

INTERVENTIONS:
Device: non-invasive cervical vagal nerve stimulation ncVNS — The ncVNS device is a rechargable, handheld device that generate a proprietary frequency-modulated electrical stimulus at low voltage (max 24V) with a max current output of 60mA. The signal consists of 1ms bursts of 5kHz sine waves repeated at 25Hz. Two stainless steel contact surfaces coated with conductive gel deliver the stimulus to the neck in the vicinity of the vagus nerve.
  Other Names: VNS
  Arms: Group 1; Group 2

SUMMARY:
More than 110,000 US Veterans living with Parkinson's disease (PD) currently receive PD-related care and services from the VA. Fall prevention is a priority for Veterans living PD. Gait disturbances are a major cause for functional dependence and the largest risk factor for falls, institutionalization, and death in PD. This SPiRE addresses the need to advance nonpharmacological rehabilitative health care of Veterans and maximizing functional outcomes by developing a non-invasive, neuromodulatory transcutaneous cervical Vagal Nerve Stimulation as an at-home intervention to improve gait and balance. This pilot clinical trial will assist with future efforts and priorities of the VA to prolong independent living and quality of life by minimizing gait and balance dysfunction experienced by Veterans living with PD.

DETAILED DESCRIPTION:
More than 110,000 US Veterans living with Parkinson's disease (PD) currently receive PD-related care and services from the VA. PD is a complex chronic neurodegenerative multisystem disorder. Fall prevention is a priority for Veterans living with PD. Gait disturbances are a major cause for functional dependence and the largest risk factor for falls, institutionalization, and death in PD. Gait abnormalities are evident at the time of PD diagnosis and are one of the most disabling features of PD. They are also difficult aspects to treat as pharmacologic agents do not address the entire spectrum of gait abnormalities. Overall management of PD symptoms can be challenging due to pharmacological interactions and drug side effects. Developing a non-pharmacological and non-invasive therapeutic to improve gait and balance is a critical need for Veterans with PD who are managing complex chronic conditions. Moreover, advancing at-home rehabilitation is ideal for a population of geriatric Veterans who are facing mobility issues, managing multiple chronic conditions and who rely on caregiver support. Non-invasive cervical Vagal Nerve Stimulation (ncVNS) may be a solution. ncVNS is currently licensed to treat and prevent migraine and other headache syndromes and is covered by the VAH for these indications. ncVNS can be self-administered, daily, at home. A hand-held device is used to make contact to the left side of the neck so that the vagal nerve is stimulated. ncVNS decreases inflammation and oxidative stress through activation of the cholinergic anti-inflammatory pathway, which in turn can contribute to gait improvements in PD. One of the most debilitating gait deficits in PD is Freezing of Gait (FOG), an episodic failure to initiate or maintain walking, especially while turning. Given that FOG, along with falls, is related to cholinergic dysfunction, both might be reduced following ncVNS. Exciting, but limited research over the past decade indicates this neuromodulatory approach has the potential to improve gait features in PD. The objectives of this SPiRE are to develop a framework for an at-home ncVNS intervention, develop an appropriate control intervention for a future larger study and gather preliminary clinical outcome data on PD-specific features. The central hypotheses are that (i) a 4 week at-home active ncVNS intervention and a sham ncVNS control condition will be acceptable and feasible to complete and (ii) active ncVNS compared to both control ncVNS and treatment as usual (TAU), will lead to greater improvements in gait, FOG, balance and fall frequency. The proposed study is a pilot, prospective parallel group randomized control trial (RCT). Twenty participants will be randomized to 4 weeks of either active (n=10) or sham ncVNS (n=10). A third group (n=10) will not receive ncVNS but will continue with their treatment as usual (TAU). The investigators will examine acute, cumulative, and sustainable effects of ncVNS. Advancing non-pharmacologic treatments to improve gait dynamics is a critical need for Veterans with PD. Moreover, advancing at-home rehabilitation is ideal for a population of geriatric Veterans who are facing multiple issues including mobility. This SPiRE is strongly aligned with VA priorities to advance rehabilitative health care of Veterans and restore their physical function to improve QoL. If the aims are achieved, the investigators will have completed necessary first steps towards developing an at-home easy to use, neuromodulatory intervention that should translate to improved gait and balance and contribute to fewer falls. This project will yield preliminary data to support a VA Merit and move forward not only the field of noninvasive and nonpharmacological interventions for PD rehabilitation but also the general field of gait and balance rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease, as diagnosis by a VA neurologist
* HY stages 2-3
* Self-report Freezing of Gait
* Able to ambulate for 2-min without an assistive device
* Parkinson's disease medications are stable for 4-weeks and expected to be on stable medications for duration of the study

Exclusion Criteria:

* Lack of decision-making capacity
* Prescribed centrally acting anticholinergics (e.g., amitriptyline) or cholinesterase inhibitors
* Musculoskeletal or additional neurological conditions that negatively impact gait and balance
* Spine or LE surgery within the past year
* Known or suspected:

  * severe atherosclerotic cardiovascular disease
  * severe carotid artery disease
  * congestive heart failure
  * known severe coronary artery disease or prior myocardial infarction
* Abnormal baseline electrocardiogram within last year
* Previous vagotomy
* Implanted metal cervical spine hardware, other metallic implants or implantable medical devices such as DBS
* History of syncope or seizures (within the last 2 years)

Ages: 50 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Stride Length | baseline and 4 weeks
  Quantitative gait analysis will be performed during a 15-meter instrumented 2-min walk test (2MWT) using the APDM Mobility Lab

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L. Kletzel, PhD BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No